CLINICAL TRIAL: NCT06125548
Title: The Effect of Lactation Management Model-Based Care Provided to Mothers With Babies in the Intensive Care Unit on the Amount of Breast Milk and Breastfeeding Duration
Brief Title: Care Based on the Lactation Management Model Provided to Mothers With Babies in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Aslı EKER, Dr, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Mersin University Midwifery
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Amount of Breast Milk
Keywords: Breastfeeding; Lactation Management Model; Breast Milk; Neonatal Intensive Care
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE RANDOMIZED CONTROLLED STUDY
Who Masked: Participant, Outcomes Assessor
Masking Description: All mothers included in the sample were assigned to experimental and control groups using the randomization table.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactation Management Model-Experimental (Experimental): The women in the experimental group were told about the care technique in accordance with the Lactation Management Model and were asked to apply it regularly for 3 days.The content of the Lactation Management Model includes skin-to-skin contact, hot application to the breast, relaxation and breast massage, and process monitoring.In this regard, the mother should apply skin-to-skin contact to her baby 12 times a day, 8 times on the 2nd day, 4 times on the 3rd day, hot application to the breast (5 minutes), relaxation technique (3 minutes) and breast massage (5 minutes manual milking, 2 minutes . nipple stimulation, stroking for 3 minutes).
  Interventions: Other: Lactation Management Model
- Non-application group- Control (No Intervention): No treatment was performed on women in the control group.

INTERVENTIONS:
Other: Lactation Management Model — The mother provides skin-to-skin contact to her baby 12 times a day, 8 times on the 2nd day, 4 times on the 3rd day, hot application to the breast (5 minutes), relaxation technique (3 minutes) and breast massage (5 minutes by hand milking, 2 minutes by breast massage). Head stimulation, stroking for 3 minutes) were asked.
  Arms: Lactation Management Model-Experimental

SUMMARY:
Using breast stimulating techniques (skin-to-skin contact, relaxation exercises, breast massage, nipple stimulation, hot application, etc.) stimulates the secretion of milk and increases its amount. This study aimed to determine the effect of care based on the lactation management model offered to mothers whose babies are in the neonatal intensive care unit, on the amount of breast milk and duration of breastfeeding.

DETAILED DESCRIPTION:
Support of prolactin and oxytocin hormones is needed for adequate production and secretion of breast milk. Many factors affect the levels of oxytocin and prolactin in the blood, such as the health status of the mother and the baby after birth, their separation for a while, nutrition, light, stress, fear, and lack of social support. Using breast stimulating techniques (skin-to-skin contact, relaxation exercises, breast massage, nipple stimulation, hot application, etc.) stimulates the secretion of milk and increases its amount. This study aimed to determine the effect of care based on the lactation management model offered to mothers whose babies are in the neonatal intensive care unit, on the amount of breast milk and duration of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,
* The baby is still in intensive care,
* Gave birth at 34 weeks of gestation and above,
* The baby was taken to intensive care within the first 3 days after birth,
* The baby will stay in the neonatal intensive care unit for at least 3 more days,
* The baby has started breastfeeding,
* Giving breast milk to the baby by expressing it,
* Not using any medication that will affect milk quantity,
* Does not have a psychiatric disease that will affect breastfeeding in the postpartum period,
* Availability by phone, language, etc. Mothers who do not have communication problems.

Exclusion Criteria:

* Not between the ages of 18-35,
* The baby is discharged from intensive care,
* Those whose gestational age is less than 34 weeks,
* The baby is taken to intensive care after the first 3 days after birth,
* The baby is in the neonatal intensive care unit for at least 3 days,
* The baby has not started breastfeeding,
* Breastfeeding,
* Those who use medication that will affect the amount of milk,
* Having a psychiatric disease that will affect breastfeeding in the postpartum period,
* Mothers with communication problems.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since it was a study on breastfeeding and breast milk, only women were included in the study.
Enrollment: 80 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Scoring system for the amount of breast milk the baby receives | Change from before implementation and 4th week of practice
  The form developed to evaluate the amount of breast milk the baby receives consists of 5 sections: urine amount, breast condition, stool amount, weight and satisfaction. Each section is grouped into 3 groups in terms of its features and is evaluated over 0, 1, 2 points. In the evaluation, 10 points mean that breast milk is received in the best way, and 7 points and below mean that breast milk is inadequate.

SECONDARY OUTCOMES:
Breast Milk and Breastfeeding Monitoring Form | Change from before implementation and 4th week of practice
  It is a form consisting of 5 questions about breastfeeding (2 questions), breast milk (2 questions) and baby's weight (1 question), developed by the researcher in line with the literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No